CLINICAL TRIAL: NCT01717768
Title: A Phase 2, Randomized, Double-blind, Dose Response Study of Oral Testosterone in Subjects With Hypogonadism
Brief Title: Oral Testosterone for the Treatment of Hypogonadism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TesoRx Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TT-002
Record Dates: First submitted 2012-10-25; First posted 2012-10-30 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Hypogonadism
Keywords: hypogonadism; Gonadal Disorders; Endocrine System Diseases; Testosterone; Testosterone enanthate; Testosterone undecanoate; Testosterone 17 beta-cypionate; Methyltestosterone; Androgens; Hormones; Hormones, Hormone Substitutes, and Hormone Antagonists; Physiological Effects of Drugs; Pharmacologic Actions; Therapeutic Uses; Anabolic Agents
MeSH Terms: conditions — Hypogonadism; Gonadal Disorders; Endocrine System Diseases | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Part 1: 120 mg BID (Experimental): Oral TSX-002 120 mg BID (total dose = 240 mg/day) for a duration of 15 days
  Interventions: Drug: TSX-002
- Part 1: 240 mg BID (Experimental): Oral TSX-002 240 mg BID (total dose = 480 mg/day) for a duration of 15 days
  Interventions: Drug: TSX-002
- Part 2: 120 mg BID (Experimental): Single cohort, open-label, nonrandomized oral TSX 002 120 mg BID (total dose = 240 mg/day) for a duration of 15 days
  Interventions: Drug: TSX-002
- Part 3: A-B-C 120 mg QD (Experimental): Open-label, randomized, 3-way crossover of 3 treatments, A, B, and C.
  * Treatment A: Oral TSX-002 (1 x 120-mg capsules) administered 30 minutes after a high-calorie, high-fat meal. No food was allowed 4 hours before the high calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  * Treatment B: Oral TSX-002 (1 x 120-mg capsules) administered 4 hours after a high-calorie, high fat meal. No food was allowed 4 hours before the high calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  * Treatment C: Oral TSX-002 (1 x 120-mg capsules) administered 30 minutes before a high-calorie, high-fat meal. No food was allowed 4 hours before the high-calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  Interventions: Drug: TSX-002
- Part 3: B-C-A 120 mg QD (Experimental): Open-label, randomized, 3-way crossover of 3 treatments, A, B, and C.
  * Treatment A: Oral TSX-002 (1 x 120-mg capsules) administered 30 minutes after a high-calorie, high-fat meal. No food was allowed 4 hours before the high calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  * Treatment B: Oral TSX-002 (1 x 120-mg capsules) administered 4 hours after a high-calorie, high fat meal. No food was allowed 4 hours before the high calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  * Treatment C: Oral TSX-002 (1 x 120-mg capsules) administered 30 minutes before a high-calorie, high-fat meal. No food was allowed 4 hours before the high-calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  Interventions: Drug: TSX-002
- Part 3: C-A-B 120 mg QD (Experimental): Open-label, randomized, 3-way crossover of 3 treatments, A, B, and C.
  * Treatment A: Oral TSX-002 (1 x 120-mg capsules) administered 30 minutes after a high-calorie, high-fat meal. No food was allowed 4 hours before the high calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  * Treatment B: Oral TSX-002 (1 x 120-mg capsules) administered 4 hours after a high-calorie, high fat meal. No food was allowed 4 hours before the high calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  * Treatment C: Oral TSX-002 (1 x 120-mg capsules) administered 30 minutes before a high-calorie, high-fat meal. No food was allowed 4 hours before the high-calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  Interventions: Drug: TSX-002
- Part 4 Cohort 1: 60 mg BID/ 60 mg TID (Experimental): Oral TSX-002 60 mg BID for 15 days then 60 mg TID for 15 days
  Interventions: Drug: TSX-002
- Part 4 Cohort 2: 90 mg BID/ 90 mg TID (Experimental): Oral TSX-002 90 mg BID for 15 days then 90 mg TID for 15 days
  Interventions: Drug: TSX-002
- Part 4 Cohort 3: 180 mg QD (Experimental): Oral TSX-002 180 mg once daily (QD) for 15 days
  Interventions: Drug: TSX-002
- Part 4 Cohort 4: 120 mg BID (Experimental): Oral TSX-002 120 mg BID for 15 days
  Interventions: Drug: TSX-002

INTERVENTIONS:
Drug: TSX-002 — TSX-002 are capsules with testosterone as the active ingredient.
  Other Names: Testosterone

SUMMARY:
Low testosterone is a condition that occurs when the body is unable to produce sufficient quantities of testosterone. The medical name for low testosterone is hypogonadism. Hypogonadism can be caused by many factors. Symptoms include: decrease in libido, lack of energy and mood swings. The goal of testosterone replacement therapy is to return testosterone levels to the normal range and relieve symptoms.

The purpose of this study is to evaluate the ability of TSX-002, which is testosterone provided in easy to swallow capsules, to maintain serum (blood) testosterone levels within the normal range in hypogonadal men. This will be determined by blood sampling at specified times during the study. The study is also intended to evaluate the tolerability of TSX-002, which will be taken orally twice per day for 15 days. In addition, the study is intended to determine a dosing regimen(s) that achieves testosterone levels within the normal range. Related Outcome Measures will be reported for Parts 1, 2, and 4.

A portion of the study (Part 3) to also assess the effect of a high-calorie, high-fat meal on the single dose pharmacokinetic exposure of TSX-002. Related outcome measures to be reported for Part 3.

ELIGIBILITY:
Inclusion Criteria:

* Prior documentation of a diagnosis of hypogonadism as evidenced by a screening serum testosterone < 300 ng/dL (based on the average of 2 morning samples taken at least 1 week apart)
* Men over the age of 18 years with a body mass index (BMI) < 39.0 kg/m2 and weighing ≥ 55 kg
* Hemoglobin levels at screening and baseline > 12.5 g/dL
* Testosterone treatment not contraindicated
* No evidence of suspected reversible hypogonadism
* Willing to abstain from current treatment for hypogonadism in accordance with approved labeling to facilitate an appropriate washout period before study participation (for nondepot formulations of testosterone only)
* Understands the requirements of the study and voluntarily consents to participate in the study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kowalczyk, DO, FACOS, Principal Investigator — Urology Group of Southern California
Locations (1):
- Urology Group of Southern California, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 130 subjects were recruited at 1 center in the US from October 2012 to May 2014. The study was designed with 4 parts, including 9 different dosages of the investigational drug.
Groups:
- Part 3: A-B-C 120 mg QD: Open-label, randomized, 3-way crossover of 3 treatments, A, B, and C.
  * Treatment A: Oral TSX-002 (1 x 120-mg capsules) administered 30 minutes after a high-calorie, high-fat meal. No food was allowed 4 hours before the high calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  * Treatment B: Oral TSX-002 (1 x 120-mg capsules) administered 4 hours after a high-calorie, high fat meal. No food was allowed 4 hours before the high calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  * Treatment C: Oral TSX-002 (1 x 120-mg capsules) administered 30 minutes before a high-calorie, high-fat meal. No food was allowed 4 hours before the high-calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  TSX-002: TSX-002 are capsules with testosterone as the active ingredient.
- Part 4 Cohort 1: 60 mg BID: Oral TSX-002 60 mg BID for 15 days
  TSX-002: TSX-002 are capsules with testosterone as the active ingredient.
- Part 4 Cohort 1: 60 mg TID: Oral TSX-002 60 mg TID for 15 days
  TSX-002 are capsules with testosterone as the active ingredient.
- Part 4 Cohort 2: 90 mg BID: Oral TSX-002 90 mg BID for 15 days
  TSX-002: TSX-002 are capsules with testosterone as the active ingredient.
- Part 4 Cohort 2: 90 mg TID: Oral TSX-002 90 mg TID for 15 days
Period: Part 1 (Duration of 15 Days)
Arm/Group | Part 1: 120 mg BID | Part 1: 240 mg BID | Part 2: 120 mg BID | Part 3: A-B-C 120 mg QD | Part 3: B-C-A 120 mg QD | Part 3: C-A-B 120 mg QD | Part 4 Cohort 1: 60 mg BID | Part 4 Cohort 1: 60 mg TID | Part 4 Cohort 2: 90 mg BID | Part 4 Cohort 2: 90 mg TID | Part 4 Cohort 3: 180 mg QD | Part 4 Cohort 4: 120 mg BID
Started | 17 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 17 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Duration of 15 Days)
Arm/Group | Part 1: 120 mg BID | Part 1: 240 mg BID | Part 2: 120 mg BID | Part 3: A-B-C 120 mg QD | Part 3: B-C-A 120 mg QD | Part 3: C-A-B 120 mg QD | Part 4 Cohort 1: 60 mg BID | Part 4 Cohort 1: 60 mg TID | Part 4 Cohort 2: 90 mg BID | Part 4 Cohort 2: 90 mg TID | Part 4 Cohort 3: 180 mg QD | Part 4 Cohort 4: 120 mg BID
Started | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3 - Treatment 1 (Duration of 1 Day)
Arm/Group | Part 1: 120 mg BID | Part 1: 240 mg BID | Part 2: 120 mg BID | Part 3: A-B-C 120 mg QD | Part 3: B-C-A 120 mg QD | Part 3: C-A-B 120 mg QD | Part 4 Cohort 1: 60 mg BID | Part 4 Cohort 1: 60 mg TID | Part 4 Cohort 2: 90 mg BID | Part 4 Cohort 2: 90 mg TID | Part 4 Cohort 3: 180 mg QD | Part 4 Cohort 4: 120 mg BID
Started | 0 | 0 | 0 | 4 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 4 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3 - Treatment 2 (Duration of 1 Day)
Arm/Group | Part 1: 120 mg BID | Part 1: 240 mg BID | Part 2: 120 mg BID | Part 3: A-B-C 120 mg QD | Part 3: B-C-A 120 mg QD | Part 3: C-A-B 120 mg QD | Part 4 Cohort 1: 60 mg BID | Part 4 Cohort 1: 60 mg TID | Part 4 Cohort 2: 90 mg BID | Part 4 Cohort 2: 90 mg TID | Part 4 Cohort 3: 180 mg QD | Part 4 Cohort 4: 120 mg BID
Started | 0 | 0 | 0 | 4 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 4 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3 - Treatment 3 (Duration of 1 Day)
Arm/Group | Part 1: 120 mg BID | Part 1: 240 mg BID | Part 2: 120 mg BID | Part 3: A-B-C 120 mg QD | Part 3: B-C-A 120 mg QD | Part 3: C-A-B 120 mg QD | Part 4 Cohort 1: 60 mg BID | Part 4 Cohort 1: 60 mg TID | Part 4 Cohort 2: 90 mg BID | Part 4 Cohort 2: 90 mg TID | Part 4 Cohort 3: 180 mg QD | Part 4 Cohort 4: 120 mg BID
Started | 0 | 0 | 0 | 4 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 4 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 4-Treatment 1 (Duration of 15 Days)
Arm/Group | Part 1: 120 mg BID | Part 1: 240 mg BID | Part 2: 120 mg BID | Part 3: A-B-C 120 mg QD | Part 3: B-C-A 120 mg QD | Part 3: C-A-B 120 mg QD | Part 4 Cohort 1: 60 mg BID | Part 4 Cohort 1: 60 mg TID | Part 4 Cohort 2: 90 mg BID | Part 4 Cohort 2: 90 mg TID | Part 4 Cohort 3: 180 mg QD | Part 4 Cohort 4: 120 mg BID
Started | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 16 | 0 | 16 | 16
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 16 | 0 | 16 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Part 4-Treatment 2 (Duration of 15 Days)
Arm/Group | Part 1: 120 mg BID | Part 1: 240 mg BID | Part 2: 120 mg BID | Part 3: A-B-C 120 mg QD | Part 3: B-C-A 120 mg QD | Part 3: C-A-B 120 mg QD | Part 4 Cohort 1: 60 mg BID | Part 4 Cohort 1: 60 mg TID | Part 4 Cohort 2: 90 mg BID | Part 4 Cohort 2: 90 mg TID | Part 4 Cohort 3: 180 mg QD | Part 4 Cohort 4: 120 mg BID
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 16 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 0 | 15 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 3: B-C-A 120 mg QD; Part 3: C-A-B 120 mg QD: Open-label, randomized, 3-way crossover of 3 treatments, A, B, and C.
  * Treatment A: Oral TSX-002 (1 x 120-mg capsules) administered 30 minutes after a high-calorie, high-fat meal. No food was allowed 4 hours before the high calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  * Treatment B: Oral TSX-002 (1 x 120-mg capsules) administered 4 hours after a high-calorie, high fat meal. No food was allowed 4 hours before the high calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  * Treatment C: Oral TSX-002 (1 x 120-mg capsules) administered 30 minutes before a high-calorie, high-fat meal. No food was allowed 4 hours before the high-calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
  TSX-002: TSX-002 are capsules with testosterone as the active ingredient.
- Total: Total of all reporting groups
Arm/Group | Part 1: 120 mg BID | Part 1: 240 mg BID | Part 2: 120 mg BID | Part 3: A-B-C 120 mg QD | Part 3: B-C-A 120 mg QD | Part 3: C-A-B 120 mg QD | Part 4 Cohort 1: 60 mg BID/ 60 mg TID | Part 4 Cohort 2: 90 mg BID/ 90 mg TID | Part 4 Cohort 3: 180 mg QD | Part 4 Cohort 4: 120 mg BID | Total
Number analyzed (Participants) | 17 | 17 | 17 | 4 | 5 | 5 | 17 | 16 | 16 | 16 | 130
Age, Customized [Number; unit: participants]
  <50 years | 2 | 4 | 8 | 1 | 1 | 0 | 4 | 4 | 9 | 5 | 38
  50-64 years | 11 | 11 | 5 | 1 | 4 | 4 | 9 | 8 | 7 | 9 | 69
  65-74 years | 3 | 2 | 3 | 1 | 0 | 1 | 3 | 4 | 0 | 2 | 19
  75 years or older | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 4
Sex/Gender, Customized [Number; unit: participants]
  Male | 17 | 17 | 17 | 4 | 5 | 5 | 17 | 16 | 16 | 16 | 130
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Black or African American | 3 | 5 | 0 | 1 | 3 | 3 | 4 | 4 | 3 | 1 | 27
  White | 13 | 12 | 17 | 3 | 2 | 2 | 10 | 12 | 13 | 12 | 96
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 17 | 4 | 5 | 5 | 17 | 16 | 16 | 16 | 130

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving a 24 Hour Average Total Serum Testosterone Concentration (Cavg,0-24h) in the Range of 300 to 1050 ng/dL After 15 Days of Treatment With TSX-002
Description: Percentage of subjects achieving a 24-hour average total serum testosterone concentration (Cavg,0-24h) in the range of 300 to 1050 ng/dL after 15 days of treatment with TSX-002. PK samples taken at 0 ,2 ,4, 5 ,6, 7, 9, 12, 14, 16, 17, 18, 21, 24 hours post-dose after 15 days of treatment for Part 1. PK samples taken at 0, 1, 2, 3, 4, 5, 6, 8, 12, 16, 17, 18, 19, 20, 21, 22, 24 hours post-dose after 15 days of treatment for Part 2. PK samples taken at 0, 1, 2, 3, 4, 5, 6, 8 ,12, 13, 14, 15, 16, 17, 18, 20, 24 hours post-dose after 15 days of treatment for Part 4.
Time Frame: 15 days
Population: All efficacy analyses were conducted based on the modified intent-to-treat (MITT) analysis population, comprised of all randomized subjects who receive at least 1 dose of study drug and have at least 1 post-baseline measurement of total serum testosterone.
Measure: Number; unit: percentage of participants
Groups:
- Part 4 Cohort 1: 60 mg TID: Oral TSX-002 60 mg three times daily (TID) for 15 days
- Part 4 Cohort 2: 90 mg TID: Oral TSX-002 90 mg TID for 15 days
  TSX-002: TSX-002 are capsules with testosterone as the active ingredient.
Arm/Group | Part 1: 120 mg BID | Part 1: 240 mg BID | Part 2: 120 mg BID | Part 4 Cohort 1: 60 mg BID | Part 4 Cohort 1: 60 mg TID | Part 4 Cohort 2: 90 mg BID | Part 4 Cohort 2: 90 mg TID | Part 4 Cohort 3: 180 mg QD | Part 4 Cohort 4: 120 mg BID
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 17 | 16 | 16 | 16 | 16
percentage of participants | 59 | 31 | 35 | 41 | 53 | 19 | 20 | 31 | 27

2. Secondary Outcome: Percentage of Subjects With Cmax ≤ 1500 ng/dL After 15 Days of Treatment 2. Percentage of Subjects With Cmax ≥ 1800 and ≤ 2500 ng/dL After 15 Days of BID Treatment 3. Percentage of Subjects With Cmax > 2500 ng/dL After 15 Days of BID Treatment
Description: Cmax. PK samples taken at 0, 2, 4, 5, 6, 7, 9, 12, 14, 16, 17, 18, 21, 24 hours post-dose after 15 days of treatment for Part 1. PK samples taken at 0, 1, 2, 3, 4, 5, 6, 8, 12, 16, 17, 18, 19, 20, 21, 22, 24 hours post-dose after 15 days of treatment for Part 2. PK samples taken at 0, 1, 2, 3, 4, 5, 6, 8, 12, 13, 14, 15, 16, 17,18, 20, 24 hours post-dose after 15 days of treatment for Part 4.
Time Frame: 15 days
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Part 1: 120 mg BID | Part 1: 240 mg BID | Part 2: 120 mg BID | Part 4 Cohort 1: 60 mg BID | Part 4 Cohort 1: 60 mg TID | Part 4 Cohort 2: 90 mg BID | Part 4 Cohort 2: 90 mg TID | Part 4 Cohort 3: 180 mg QD | Part 4 Cohort 4: 120 mg BID
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 17 | 16 | 16 | 16 | 16
percentage of subjects
  Percentage of subjects with Cmax ≤ 1500 ng/dL afte | 100 | 100 | 94.1 | 100 | 100 | 100 | 100 | 100 | 93.75
  Percentage of subjects with Cmax ≥ 1800 and ≤ 2500 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6.25
  Percentage of subjects with Cmax > 2500 ng/dL afte | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Other Pre Specified Outcome: Cavg 0-24 Hrs (ng/dL) After 120 mg Dose
Description: PK samples taken at 0, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24 hours post-dose after 1 day of treatment for Part 3. Mean of Cavg values from all time points for 14 subjects.
Time Frame: 24 hrs
Population: All subjects that received 120 mg TSX-002 under defined Treatment conditions (timing of high-calorie, high-fat meal).
Measure: Least Squares Mean (Standard Deviation); unit: ng/dL
Groups:
- Part 3:120 mg QD Treatment A: Treatment A: Oral TSX-002 (1 x 120-mg capsules) administered 30 minutes after a high-calorie, high-fat meal. No food was allowed 4 hours before the high calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
- Part 3:120 mg QD Treatment B: Treatment B: Oral TSX-002 (1 x 120-mg capsules) administered 4 hours after a high-calorie, high fat meal. No food was allowed 4 hours before the high calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
- Part 3:120 mg QD Treatment C: Treatment C: Oral TSX-002 (1 x 120-mg capsules) administered 30 minutes before a high-calorie, high-fat meal. No food was allowed 4 hours before the high-calorie, high-fat meal and no food was allowed for at least 10 hours after dosing.
Arm/Group | Part 3:120 mg QD Treatment A | Part 3:120 mg QD Treatment B | Part 3:120 mg QD Treatment C
Number analyzed (Participants) | 14 | 14 | 14
ng/dL | 296 (108) | 297 (75) | 273 (109)

4. Other Pre Specified Outcome: AUC 0-24 Hrs After 120 mg Dose of TSX-002
Description: AUC 0-24 hrs with PK samples taken at 0, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24 hours post-dose after 1 day of treatment for Part 3.
Time Frame: 24 hrs
Population: All subjects that received 120 mg TSX-002 under defined Treatment conditions (timing of high-calorie, high-fat meal).
Measure: Median (Standard Deviation); unit: hr×ng/dL
Arm/Group | Part 3:120 mg QD Treatment A | Part 3:120 mg QD Treatment B | Part 3:120 mg QD Treatment C
Number analyzed (Participants) | 14 | 14 | 14
hr×ng/dL | 1941 (1198) | 2117 (1351) | 1516 (1217)

ADVERSE EVENTS:
Time Frame: The adverse events presented were collected from start of drug treatment to discontinuation or completion of study participation.
Groups:
- Part 4 Cohort 1: 60 mg TID: Oral TSX-002 60 mg TID for 15 days
  TSX-002: TSX-002 are capsules with testosterone as the active ingredient.
Arm/Group | Part 1: 120 mg BID | Part 1: 240 mg BID | Part 2: 120 mg BID | Part 3: A-B-C 120 mg QD | Part 3: B-C-A 120 mg QD | Part 3: C-A-B 120 mg QD | Part 4 Cohort 1: 60 mg BID | Part 4 Cohort 1: 60 mg TID | Part 4 Cohort 2: 90 mg BID | Part 4 Cohort 2: 90 mg TID | Part 4 Cohort 3: 180 mg QD | Part 4 Cohort 4: 120 mg BID
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/4 | 0/5 | 0/5 | 0/17 | 0/17 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 6/17 | 8/17 | 6/17 | 0/4 | 2/5 | 2/5 | 3/17 | 3/17 | 0/16 | 2/16 | 6/16 | 3/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: 120 mg BID (N=17) | Part 1: 240 mg BID (N=17) | Part 2: 120 mg BID (N=17) | Part 3: A-B-C 120 mg QD (N=4) | Part 3: B-C-A 120 mg QD (N=5) | Part 3: C-A-B 120 mg QD (N=5) | Part 4 Cohort 1: 60 mg BID (N=17) | Part 4 Cohort 1: 60 mg TID (N=17) | Part 4 Cohort 2: 90 mg BID (N=16) | Part 4 Cohort 2: 90 mg TID (N=16) | Part 4 Cohort 3: 180 mg QD (N=16) | Part 4 Cohort 4: 120 mg BID (N=16)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site phlebitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sluggishness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anger (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: At 60 days prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the Site shall provide to Sponsor a copy and allow Sponsor 60 days to review and comment and provide written permission prior to publication.